CLINICAL TRIAL: NCT07329673
Title: An Examination of the Performance of QbMobile in Differential Diagnosis Associated With ADHD Symptoms.
Status: Not yet recruiting | Type: Observational
Sponsor: Qbtech AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00090568 QB25-01
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Bi-Polar Disorder; Autism Spectrum Disorder (ASD); Major Depression Disorders; Separation Anxiety Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder (GAD)
MeSH Terms: conditions — Bipolar Disorder; Autism Spectrum Disorder; Anxiety, Separation; Phobia, Social; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- ASD: Eligible participants being referred for their initial assessment or have a diagnosis of ASD but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)
- Bipolar disorder: Eligible participants being referred for their initial assessment or have a diagnosis of Bipolar Disorder but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)
- MDD: Eligible participants being referred for their initial assessment or have a diagnosis of MDD but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)
- Separation Anxiety Disorder: Eligible participants being referred for their initial assessment or have a diagnosis of Separation Anxiety Disorder but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)
- Social Anxiety Disorder: Eligible participants being referred for their initial assessment or have a diagnosis of Social Anxiety Disorder but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)
- Generalized Anxiety Disorder: Eligible participants being referred for their initial assessment or have a diagnosis of Generalized Anxiety Disorder but currently not receiving treatment who are attending a clinic visit at study sites will be approached by a clinic research staff about the study or contacted prior to their appointment.
  Interventions: Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device)

INTERVENTIONS:
Device: Digital software application for cognitive performance and activity measurement (QbMobile, investigational device) — Participants will complete two non-invasive, 10-minute digital tests using the QbMobile Investigational Device-one at the clinic and one at home the following day. The tests objectively measure cognitive performance and activity levels and will not influence clinical diagnosis or treatment in this study.

SUMMARY:
The purpose of this study is to evaluate QbMobile's ability to collect objective data to identify specific symptom profiles in differential diagnoses (ASD, MDD, Bipolar Disorder and Anxiety Disorder) that are common with ADHD.

DETAILED DESCRIPTION:
This study aims to evaluate the performance of QbMobile in children, adolescents, and adults assessed for and diagnosed with ASD (Autism Spectrum Disorder, MDD (Major Depressive Disorder), Bipolar Disorder, or Anxiety Disorder, or has a prior diagnosis of one of the included disorders but is not currently receiving treatment. Participants will complete the 10-minute QbMobile test on their personal device during a scheduled clinical visit. They will then repeat the test remotely the following day at the same time as the previous test +/-3 hours. Participants will be asked to complete QbMobile prior to initiating any treatment.

Note on Outcome Measures Presentation:

The IRB-approved protocol defines endpoints broadly (e.g., identification of QbMobile domain profiles, classification accuracy, variability, and exploratory analyses). To comply with ClinicalTrials.gov requirements that each outcome measure represent a single assessment with a single unit of measure, these endpoints are operationalized into separate outcome measures corresponding to individual QbMobile metrics (domain SD-scores, Total Score [0-100], accuracy percentages, variability estimates).

This operationalization does not introduce new scientific endpoints or alter study objectives, design, or analyses. It ensures clarity and compliance for registry reporting while maintaining alignment with the approved protocol.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent (including parent/legal guardians consent when this is required for individuals under 18 years old and assent as is required based on the age of participant) for QbMobile;
* Aged > 6 years and < 60 years old;
* Referred for an initial assessment for ASD, MDD, Bipolar Disorder or Anxiety Disorder (Separation Anxiety Disorder, Social Anxiety Disorder, Generalized Anxiety Disorder (GAD)) or has a prior diagnosis of one of the included disorders but is not currently receiving treatment;
* Meets DSM-5 or ICD-11 criteria for a primary diagnosis of ASD, MDD, Bipolar Disorder or Anxiety Disorder per sites standard clinical procedures;
* Have adequate sensory and physical ability to complete QbMobile;
* Possess or have access to an iPhone model that supports QbMobile.

Exclusion Criteria:

* Intellectual disability designated by IQ<70;
* Has a DSM-5 or ICD-11 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, psychotic disorder due to another medical condition, PTSD, antisocial personality disorder, or borderline personality disorder;
* Has a primary diagnosis of ADHD (combined, inattentive, or hyperactivity/impulsive presentation);
* Has a concurrent medical diagnosis that could significantly affect test performance such as brain injuries, Parkinson's disease, current epilepsy or active seizures, amyotrophic lateral sclerosis (ALS), multiple sclerosis, dementias (e.g. vascular dementia, Alzheimer disease, etc);
* Has other conditions that could affect test performance (migraine or other types of severe headache, chronic or acute pain);
* Use of prescription medications (e.g., anxiolytics, sedative medications) taken on the day before completing QbMobile that could significantly affect performance;
* Substance use (e.g., alcohol, drugs) that may affect performance on the day of the tests.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Potential study participants who meet the eligibility criteria will be identified through referrals and recruitment efforts at the participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Identification of QbMobile Domain Profiles Using SD-Scores and Total Score (0-100) | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2)
  QbMobile is a software application that measures cognitive performance and activity levels, including attention, impulsivity, activity, and movement patterns. The study will identify statistically distinct QbMobile domain profiles for each diagnostic group (ASD, MDD, Bipolar Disorder, Anxiety Disorder) using domain SD-scores and the QbMobile Total Score (0-100). (Component metrics are listed as secondary outcomes to meet single-measure reporting requirements.)

SECONDARY OUTCOMES:
QbMobile Domain SD-Scores (Attention, Impulsivity, Activity, Movement) - Group Differences | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2)
  QbMobile is a software application that measures cognitive performance and activity levels. Domain scores will be analyzed as SD-scores to assess differences among diagnostic groups (ASD, MDD, Bipolar Disorder, Anxiety Disorder).
QbMobile Total Score (0-100) - Group Differences | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2)
  QbMobile is a software application that measures cognitive performance and activity levels. The Total Score (0-100; higher values indicate greater likelihood of ADHD symptomatology) will be compared across diagnostic groups to assess differences.
Classification Accuracy Using QbMobile Domain SD-Scores | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2)
  QbMobile is a software application that measures cognitive performance and activity levels. Classification accuracy among diagnostic groups will be evaluated using domain SD-scores; metrics will include sensitivity, specificity, and predictive values.
Classification Accuracy Using QbMobile Total Score (0-100) | QbMobile completed at Visit 1 (Day 1) and Visit 2 (Day 2)
  QbMobile is a software application that measures cognitive performance and activity levels. Classification accuracy among diagnostic groups will be evaluated using the Total Score; metrics will include sensitivity, specificity, and predictive values based on prespecified thresholds.
Comparison of QbMobile Domain SD-Scores with Normative Dataset | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2).
  QbMobile is a software application that measures cognitive performance and activity levels. Domain SD-scores will be compared with the age- and sex-adjusted normative dataset to identify differences between diagnostic groups and normative patterns.
Comparison of QbMobile Total Score (0-100) with Normative Distribution | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2).
  QbMobile is a software application that measures cognitive performance and activity levels. Total Scores will be compared with the normative distribution to identify deviations from expected values.
Variability in Differentiation Using QbMobile Domain SD-Scores | Two QbMobile tests: at the clinic (Visit 1) and remotely the following day (Visit 2).
  QbMobile is a software application that measures cognitive performance and activity levels. Variability in group differentiation will be assessed using domain SD-scores (e.g., confidence intervals and variance estimates across repeated measures).
Variability in Differentiation Using QbMobile Total Score (0-100) | QbMobile completed at Visit 1 (Day 1) and Visit 2 (Day 2).
  QbMobile is a software application that measures cognitive performance and activity levels. Variability will be assessed using Total Scores (e.g., confidence intervals and variance estimates across repeated measures).
Exploratory Analysis of Additional QbMobile Domain Parameters (SD-Based) | QbMobile completed at Visit 1 (Day 1) and Visit 2 (Day 2).
  Consistent with the protocol statement that "all data collected from QbMobile during this study will be available to explore additional domain parameters," exploratory analyses will examine QbMobile domain data using SD-based metrics to identify additional parameters for further analysis.
Exploratory Analysis of Additional QbMobile Parameters from Total Score and Raw Performance Data | Visit 1 (clinic) and Visit 2 (remote, next day).
  Consistent with the protocol statement that "all data collected from QbMobile… will be available to explore additional domain parameters," exploratory analyses will use the QbMobile Total Score (0-100) and raw performance data (e.g., response time, error counts, movement traces) to identify additional parameters for further analysis.

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the research, limited access to supporting data may be granted upon reasonable request under confidentiality agreements from the corresponding sponsor.